CLINICAL TRIAL: NCT02279953
Title: An Interventional, Randomised, Double-blind, Parallel-group, Placebo-controlled Study on the Efficacy of Vortioxetine on Cognitive Dysfunction in Patients With Partial or Full Remission of Major Depressive Disorder
Brief Title: Efficacy of Vortioxetine on Cognitive Dysfunction in Patients With Partial or Full Remission of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15905A; 2014-000229-19 (EudraCT Number)
Record Dates: First submitted 2014-10-21; First posted 2014-10-31 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vortioxetine 10-20 mg (Experimental): daily, encapsulated, orally
  Interventions: Drug: Vortioxetine 10-20 mg; Drug: Placebo
- Vortioxetine 10-20 mg + SSRI (Experimental): daily, encapsulated, orally
  Interventions: Drug: Vortioxetine 10-20 mg; Drug: SSRI
- SSRI (Experimental): licensed doses, encapsulated, orally
  Interventions: Drug: Placebo; Drug: SSRI

INTERVENTIONS:
Drug: Vortioxetine 10-20 mg
  Other Names: Brintellix®; Lu AA21004
  Arms: Vortioxetine 10-20 mg; Vortioxetine 10-20 mg + SSRI
Drug: Placebo
  Arms: SSRI; Vortioxetine 10-20 mg
Drug: SSRI — escitalopram, citalopram or sertraline
  Arms: SSRI; Vortioxetine 10-20 mg + SSRI

SUMMARY:
To assess the efficacy of vortioxetine (10 to 20 mg/day) as adjunctive treatment to stable selective serotonin reuptake inhibitor (SSRI) dose versus stable SSRI monotherapy on cognitive performance (focusing on the aspect concerning speed of processing, executive functioning and attention) in patients who are in partial or full remission from their Major Depressive Episode (MDE).

ELIGIBILITY:
Inclusion Criteria:

* The patient has achieved either partial (some symptoms of a MDE are present but full criteria are not met) or full remission of major depressive disorder (MDD), diagnosed according to DSM-IV-TR™.
* The patient has HAMD-17 total score ≤10.
* The patient has received SSRI monotherapy for the MDE from which the patient is currently in full or partial remission for ≥12 weeks at licensed doses and been on stable dose ≥8 weeks prior to Screening Visit.
* The patient has ≥50% response to current SSRI treatment (Antidepressant Treatment Response Questionnaire [ATRQ]).
* The patient has a PDQ-D total score >25.
* The patient is a man or woman, aged ≥18 and ≤65 years.

Exclusion Criteria:

* The patient has a score ≥70 on the DSST (numbers of correct symbols) at the Baseline Visit.
* The patient is, in the opinion of the investigator, not able to complete the neuropsychological tests validly at the Baseline Visit.
* The patient has physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the neuropsychological tests.
* The patient is diagnosed with reading disability (dyslexia).
* The patient has a history of lack of response to previous adequate treatment with vortioxetine.
* The patient has any current psychiatric disorder or Axis I disorder (according to DSM-IV-TR™ criteria) other than MDD, as assessed using Mini International Neuropsychiatric Interview (MINI).
* The patient has a current or has had a diagnosis of dysthymic disorder within 3 months preceding the onset of the depressive episode from which the patient is currently in full or partial remission (DSM-IV-TR™ criteria).
* The patient has borderline, schizotypal, schizoid, paranoid, histrionic, antisocial personality disorders (axis II) as comorbid or primary diagnosis (DSM-IV-TR™ criteria).
* The patient suffers from personality disorders, mental retardation, pervasive development disorder, attention-deficit/hyperactivity disorder, organic mental disorders, or mental disorders due to a general medical condition (DSM-IV-TR™ criteria).
* The patient has a current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features (DSM-IV-TR™ criteria).

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Digit Symbol Substitution Test (DSST): number of correct symbols | Baseline to Week 8

SECONDARY OUTCOMES:
Change in Rey Auditory Verbal Learning Test (RAVLT) score: memory (delayed recall) and learning [acquisition]) | Baseline to Week 8
Change in Trail Making Test (TMT) score: TMT-A; speed of processing | Baseline to Week 8
Change in TMT score: TMT-B; executive functioning | Baseline to Week 8
Change in reaction time score: Choice Reaction Time (CRT); attention | Baseline to Week 8
Change in reaction time score: Simple Reaction Time (SRT); psychomotor speed | Baseline to Week 8
Change in Stroop Colour Naming Test (STROOP): incongruent score; executive functioning | Baseline to Week 8
Change in STROOP: congruent score; speed of processing | Baseline to Week 8
Change in Perceived Deficits Questionnaire - Depression (PDQ-D) total score | Baseline to Week 8
Change in Hamilton Depression Rating Scale-17 (HAMD-17) total score | Baseline to Week 8
Change in Clinical Global Impression - Severity of Illness (CGI-S) | Baseline to Week 8
Clinical Global Impression - Global Improvement (CGI-I) score | Week 8
Change in University of San Diego Performance-based Skills Assessment - Brief (UPSA-B) total score | Baseline to Week 8
Number of adverse events | Baseline to Week 12
Columbia Suicide Severity Rating Scale (C-SSRS) categorisation based on Columbia Classification Algorithm of Suicide Assessment (C-CASA) definitions (1, 2, 3, 4 and 7) | Baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (17):
- Estonia (2):
  - EE001, Tallinn
  - EE002, Tallinn
- Finland (6):
  - FI002, Helsinki
  - FI003, Helsinki
  - FI005, Helsinki
  - FI001, Kuopio
  - FI006, Kupio
  - FI004, Turku
- Germany (5):
  - DE002, Berlin
  - DE001, Bielefeld
  - DE005, Bochum
  - DE003, Frankfurt
  - DE004, Mittweida
- Serbia (2):
  - RS002, Belgrade
  - RS001, Kragujevac
- Slovakia (2):
  - SK003, Levice
  - SK002, Rimavská Sobota

REFERENCES:
- See also: Results EudraCT 2014-000229-19 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-000229-19/results